CLINICAL TRIAL: NCT01375920
Title: Antiglucocorticoid Augmentation of antiDepressants in Depression
Acronym: ADD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jane Barnes (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Jane Barnes, Professor, Northumberland, Tyne and Wear NHS Foundation Trust
Organization: Northumberland, Tyne and Wear NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EME-08/43/39; ISRCTN (Registry Identifier: ISRCTN: 45338259); 2009-015165-31 (EudraCT Number); EME Grant (Other Grant/Funding Number: 08/43/39)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Depression
Keywords: Depression; Antiglucocorticoid; Anti-depressants
MeSH Terms: conditions — Depression | interventions — Metyrapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metyrapone, daily medication (Active Comparator): 500 milligrams Metyrapone to be taken orally twice daily for 3 weeks.
  Interventions: Drug: Metyrapone
- placebo (Placebo Comparator): a matched placebo will be given for patients to take twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metyrapone — 500 milligrams to be taken twice a day orally
  Other Names: Metyrapone also known as Metopirone
  Arms: Metyrapone, daily medication
Drug: placebo — a matched placebo will be administered to patients to take twice a day for 3 weeks
  Arms: placebo

SUMMARY:
Depression is one of the most common mental health problems, with at least one in six adults suffering from this at some time in their life. It can become long-lasting and frequently recurs. Depression has a large negative impact on quality of life of patients and their carers and it has also been shown to be one of the leading causes of working age adults receiving disability payments in the UK. The need for improved treatment has been recognised by the Department of Health and others. Improvements in drug treatments are therefore required. There has been recent increased understanding of some of the causes of the frequent lack of complete response seen with antidepressants. The stress hormone, cortisol, is often elevated or poorly controlled in depression and there is laboratory and clinical research to show that this hormonal change reduces the benefits from antidepressants with associated poor outcome and memory problems. Recently it has been shown in small studies that giving treatments that reduce cortisol or block its harmful effects for between 1 and 3 weeks overcome these negative consequences. Our group is particularly interested and experienced in this topic. The investigators plan to study a drug that decreases cortisol levels in people who have not recovered with standard antidepressants so that the investigators can find out the usefulness of this treatment (compared with placebo (dummy tablet)) in day to day life as well as checking closely for side-effects (the initial studies have shown that the particular drug the investigators wish to study (metyrapone) has few side effects). The investigators will also measure cortisol and see if its level can tell us which people do best with this treatment. The investigators will carry out this study in 3 centres across the UK. The investigators will carry out some additional tests of specific sorts of memory and decision making and also do this while scanning the brain (in a painless test). The results of these tests, along with tests of brain wave patterns, should help us understand more fully how this new treatment is working and who responds best to it. The study will help us find out if this drug should be used more widely for people not responding to standard treatments and will also lead on to the development of other new treatments with an anti-cortisol effect to help tackle the major problem of poor outcome from depression.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Depression Severity: Hamilton Depression Rating Scale (HDRS17) score ≥18, consistent with a moderate to severe episode. The stability of the patient's clinical state will also be assessed at week 0. A repeat HDRS17 score at time 0 is required ≥18 or greater.
2. Treatment refractoriness: assessed using the Massachusetts General Hospital (MGH) staging method. This defines minimum effective doses of all currently-available antidepressants and an "adequate trial" as being for at least six weeks. For the trial to be considered a "failure", it must have been considered by the clinical team to have been ineffective rather, than the drug not having been taken or tolerated. Patients must have failed to have responded to at least their second trial of an antidepressant. This equates to a minimum score of two on MGH staging. The maximum MGH score for inclusion in the study will be 10. A UK study showed mean MGH scores in primary care patients of less than one, in secondary care mental health settings of around five and of 11 in a population of patients referred to a tertiary centre (Dr D Christmas, Dundee, Personal Communication).
3. Current antidepressant treatment: patients must be taking monotherapy or combination antidepressant therapy which includes a serotonergic drug (an SSRI, a tertiary amine tricyclic, venlafaxine, duloxetine or mirtazapine). They must not be on noradrenergic antidepressant monotherapy (e.g. with lofepramine, imipramine or reboxetine). At the point of randomisation, patients must have been on their current antidepressant medication, at the current dose, for a minimum of four weeks.
4. Age: 18-65. For the mechanistic sub-studies the patients upper age limit is 60.

Healthy Control Inclusion Criteria:

1. Aged 18-60.
2. Currently psychiatrically well, confirmed through SCID interview. HDRS17 score of ≤5, and no current psychotropic medication.
3. No past history of psychiatric illness, as revealed by SCID interview, or requiring any treatment (formal psychotherapy or psychotropic medication).
4. No first degree family history of psychiatric illness.

Patient Exclusion Criteria:

1. Any other DSM IV Axis I disorder other than an anxiety disorder unless the depressive episode is considered to be secondary to the anxiety disorder, confirmed using the Structured Clinical Interview for DSM (SCID).
2. Physical co-morbidity which would render the use of Metyrapone inappropriate, including untreated hypothyroidism, disorders of steroid production, current, severe cardiac failure, current, severe or frequent angina, current renal failure or myocardial infarction within the last year.
3. Pregnancy, determined by history and, if indicated, urine pregnancy test.
4. Mothers who are breastfeeding.
5. Use of concomitant medication that would interfere, in a pharmacodynamic or pharmacokinetic manner, with Metyrapone.
6. Dependence on alcohol or other drug in the past 12 months, and/or current harmful use of alcohol or other drug.
7. Recently having taken part in another research study that could interfere with the results of this one.

Healthy Control Exclusion Criteria:

1. Any physical ill health which would render the use of Metyrapone inappropriate, including untreated hypothyroidism, disorders of steroid production, current, severe cardiac failure, current, severe or frequent angina, current renal failure, or myocardial infarction within the last year. NOTE: healthy controls are NOT treated with Metyrapone.
2. Pregnancy, determined by history and, if indicated, urine pregnancy test.
3. Mothers who are breastfeeding.
4. Use of any medication that would interfere, in a pharmacodynamic or pharmacokinetic manner, with Metyrapone.
5. Dependence on alcohol or other drug in the past 12 months, and/or current harmful use of alcohol or other drug.
6. Presence of any metal implants or foreign bodies such as from a surgical implant, accident or injury [this criteria only applies to those undergoing the fMRI scans - this is all 30 healthy subjects recruited in the North West (NW)and 15 of the 25 recruited in the North East (NE)].
7. Recently having taken part in another research study that could interfere with the results of this one.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in Montgomery-Asberg Depression Rating Scale (MADRS) from week 0 to +5 weeks. | 5 weeks
  The primary outcome will be the change in Montgomery-Asberg Depression Rating Scale (MADRS) from week 0 to +5 weeks.

SECONDARY OUTCOMES:
Secondary outcomes related to mood will be the Montgomery-Asberg Depression Rating Scale (MADRS) measured at time +3, +5, +8, +16 and + 24 weeks relative to baseline. | up to 6 months
  Secondary outcomes related to mood will be the Montgomery-Asberg Depression Rating Scale (MADRS) measured at time randomisation, +3, +5, +8, +16 and + 24 weeks relative to baseline.
Clinical Anxiety Scale (CAS) | up to 6 months
  1. Mood as measured by YMRS and BDI at time 0, +3, +5, +8, +16, +24 weeks
  2. Anxiety as measured by the CAS and STAI at time 0, +3, +5, +8, +16, +24 weeks
  3. Quality of life, assessed using the EQ-5D at weeks 0, +3, +5, +8, +16, +24
  4. Tolerability assessed using the TSES and self-report at weeks 0, +3, +5, +8 (additional self-report at weeks +1, +2 and +4)
  5. Suicide risk assessed at weeks 0, +1, +3, +5, +8, +16, +24
  6. Hypothalamic-Pituitary-Adrenal (HPA) axis function assessed by salivary cortisol awakening response (CAR) and sample at 11 pm at weeks 0, +3 and +5
  7. Safety assessments including blood pressure, urea and electrolytes and plasma cortisol levels at weeks -2, +1 and +5
Quality of life will be assessed using the self-completed EuroQol EQ-5D instrument (http://www.euroqol.org/). The EQ-5D will be completed at 0, +3, +5, +8, +16 and + 24, weeks. | up to 6 months
  Quality of life will be assessed using the self-completed EuroQol EQ-5D instrument (http://www.euroqol.org/). The EQ-5D will be completed at 0, +3, +5, +8, +16 and + 24, weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ian N Ferrier, MRCPsych, Study Chair — Newcastle University; Richard H McAllister-Williams, FRCP, Principal Investigator — Newcastle University; Stuart Watson, MRCPsych, Principal Investigator — Newcastle University; Ian M Anderson, FRCPsych, Principal Investigator — Manchester University; Allan O House, MRCPsych, Principal Investigator — Leeds University; Elaine M McColl, PhD, Study Director — Newcastle University; Ian N Steen, PhD, Study Director — Newcastle University; Heinz CR Grunze, BoardCertPsy, Principal Investigator — Newcastle University; Peter M Haddad, MRCPsych, Principal Investigator — Manchester University; Thomas A Hughes, MRCPsych, Principal Investigator — Leeds Partnerships NHS Foundation Trust; Adrian Lloyd, MRCPsych, Principal Investigator — Northumberland, Tyne and Wear NHS Trust; Andrew M Blamire, BSc, PhD, Principal Investigator — Newcastle University
Locations (11):
- United Kingdom (11):
  - Stockton Affective Disorders Service, Newcastle upon Tyne, Teesside
  - Newcastle Community Mental Health Team, Newcastle upon Tyne, Tyne and Wear
  - Regional Affective Disorders Service, Newcastle upon Tyne, Tyne and Wear
  - North Tyneside Community Mental Health Team, Newcastle upon Tyne, Tyne and Wear
  - Newcastle Magnetic Resonance Centre, Newcastle upon Tyne, Tyne and Wear
  - Bradford District Care Trust, Bradford
  - Leeds Community Mental Health Team, Leeds
  - Affective Disorders Service, Manchester
  - Manchester Community Mental Health Team, Manchester
  - Manchester Magnetic Resonance Centre, Manchester
  - Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne